CLINICAL TRIAL: NCT06562023
Title: Botulinum Toxin Versus Mesotherapy on Enhancement of Facial Scarring (A Randomized Controlled Clinical Trial)
Brief Title: Botulinum Toxin and Mesotherapy on Enhancement of Facial Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0926-5/2024
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Facial Scars
MeSH Terms: interventions — Botulinum Toxins, Type A; Mesotherapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BTA injection (Experimental)
  Interventions: Other: Botulinum Toxin Type A
- Mesotherapy (Experimental)
  Interventions: Other: Mesotherapy
- Control (No Intervention)

INTERVENTIONS:
Other: Botulinum Toxin Type A — Patients will receive BTA injection within a period of 5 days after primary closure.
  Arms: BTA injection
Other: Mesotherapy — Patients will receive mesotherapy growth factor serum with a derma pen within a period of 5 days after primary closure.
  Arms: Mesotherapy

SUMMARY:
Most of the body's tissues can undergo wound repair following a disruption of tissue integrity. Upon healing, these wounds result in scar formation. The scars widen when the overlying musculature pulls apart suture lines. Botulinum Toxin A (BTA) is known to prevent fibroblast proliferation and it also induces temporary muscle paralysis. Also, mesotherapy is the non-invasive transdermal injection which can aid the skin to increase collagen and elastin production. Thus, both techniques are eligible for enhancement of facial scars.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from vertical or oblique forehead lacerations caused by trauma.
* Recent and fresh wounds.
* Atrophic scar (linear scar).

Exclusion Criteria:

* Infected wound.
* Patient on chemotherapy treatment and history of malignancy.
* Patients suffering from burns on the forehead or complicated lacerations.
* Allergy to drugs used in this study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-11-19 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Change in scar appearance | Baseline, 1 month, 3 months, 6 months
  The Vancouver Scar Scale (VSS) will be measured to calculate scar appearance. The VSS evaluates four indicators: vascularity, pigmentation, pliability, and height. It has a score ranging from 0-13.
  * Vascularity: Normal 0, Pink 1, Red 2, Purple 3
  * Pigmentation: Normal 0, Hypopigmentation 1, Hyperpigmentation 2
  * Pliability: Normal 0, Supple 1, Yielding 2, Firm 3, Ropes 4, Contracture 5
  * Height: Flat (0), < 2 mm (1), 2-5 mm (2), > 5 mm (3)
Change in wound width | Baseline, 1 month, 3 months, 6 months
  The mean wound width will be measured using a graduated Vernier caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt